CLINICAL TRIAL: NCT04658927
Title: Intracanalicular Dexamethasone Used in Conjunction With ILUX for the Treatment of Meibomian Gland Dysfunction (MGD) in Patients With Evaporative Dry Eye and Evidence of Clinically Significant Inflammation.
Brief Title: Dextenza With ILUX for Treatment of MGD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Warrenville Eyecare (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIJM Study
Record Dates: First submitted 2020-11-18; First posted 2020-12-09 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Meibomian Gland Dysfunction; Evaporative Dry Eye
Keywords: dry eye; meibomian gland dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes | interventions — Dexamethasone; Calcium Dobesilate; Prednisone

STUDY DESIGN:
Intervention Model Description: All eyes will undergo iLUX MGD Treatment System for the treatment of evaporative DED secondary to MGD. Patients will have their most symptomatic eye selected to receive the dexamethasone intracanalicular insert at the day of the iLUX MGD Treatment System (study eye). There will be 2 groups:
  Group 1: fellow eye will receive topical prednisolone acetate 1% on a 4,3,2,1 taper for 30 days (control eye) Group 2: fellow eye will receive punctal "sham" dilation (control eye).
  If there is no obvious symptomatic difference, the right eye will receive the intracanalicular insert.
  Screening Visit Treatment Visit 1 week follow up
  1 month follow up 3 month follow up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dexamethosone intracanalicular insert (Experimental): All 30 eyes will undergo iLUX MGD Treatment System for the treatment of evaporative DED secondary to MGD. Patients will have their most symptomatic eye selected to receive the dexamethasone intracanalicular insert at the day of the iLUX MGD Treatment System (study eye).
  Interventions: Drug: Dexamethasone, 0.4mg
- Group 1: Prednisolone actetate 1% (Active Comparator): 15 fellow eye will undergo iLux and receive topical prednisolone acetate 1% on a 4,3,2,1 taper for 30 days.
  Interventions: Drug: Prednisone acetate
- Group 2: Sham dilation (Sham Comparator): 15 fellow eye will undergo ILux and receive punctal "sham" dilation (control eye).
  Interventions: Other: Control

INTERVENTIONS:
Drug: Dexamethasone, 0.4mg — iLUX + dextenza
  Other Names: dextenza
  Arms: Dexamethosone intracanalicular insert
Drug: Prednisone acetate — Prednisolone acetate 1% and iLux
  Arms: Group 1: Prednisolone actetate 1%
Other: Control — iLUX alone.
  Arms: Group 2: Sham dilation

SUMMARY:
To evaluate the benefit of treatment with a physician administered intracanalicular dexamethasone insert in evaporative dry eye disease (DED) patients with meibomian gland disfunction (MGD) and underlying inflammation undergoing iLUX MGD Treatment System.

DETAILED DESCRIPTION:
This prospective study will use a fellow-eye design for 30 participants, (2 groups of 15) equating to 60 eyes. All eyes will receive bilateral iLUX MGD Treatment System. The most symptomatic eye will be selected to receive DEXTENZA® insertion on the day of the procedure (study eye). In group 1, the other eye will be assigned to receive prednisolone acetate 1% on a 4,3,2,1 month taper schedule (active comparator). In group 2, the other eye will receive punctal "sham" dilation (control eye). If there is no obvious symptomatic difference, the right eye will receive the intracanalicular insert. The study group will consist of 30 eyes receiving DEXTENZA® insertion. The control group will consist of 15 eyes receiving prednisolone acetate 1% and 15 eyes receiving sham punctum dilation. Thus, for every eye in the study group, there will be a paired eye with similar baseline characteristics in the control group sourced from the same participant. This fellow-eye design allows for greater control of potential confounders tied to participants' systemic and ocular health.

ELIGIBILITY:
Inclusion Criteria:

* A patient's study eye must meet the following criteria to be eligible for inclusion in the study:

  * 18 years of age or older
  * Evaporative DED with MGD and clinically significant inflammation
  * Willing and able to comply with clinic visits and study related procedures
  * Willing and able to sign the informed consent form

Exclusion Criteria:

* A patient who meets any of the following criteria will be excluded from the study:

  * Patients under the age of 18.
  * Pregnancy (must be ruled out in women of child-bearing age with pregnancy test)
  * Active infectious systemic disease
  * Active infectious ocular or extraocular disease
  * Altered nasolacrimal flow of either acquired, induced, or congenital origin
  * Hypersensitivity to dexamethasone
  * Patient being treated with either topical, oral, or intravenous steroids
  * Patients with severe disease that warrants critical attention, deemed unsafe for the study by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Change in Meibomian gland score (MGS) | Assessed on week 1, week 4 and week 12.
  Change from baseline in meibomian gland scores (expressibility and quality)
Patient satisfaction with treatment | Assessed on week 12
  preference for therapy as measured by COMTOL

SECONDARY OUTCOMES:
Change in Matrix metalloproteinase (MMP) -9 | Assessed on Week 1, 4, 12
  Mean change in MMP-9 from baseline as measured by InflammaDry
Change in corneal staining | Assessed on week 1, week 4 and week 12
  Mean change in ocular surface staining (sodium fluorescein and lissamine green) from baseline as measured by the National Eye Institute grading scale
Change in tear osmolarity | Assessed on week 1, week 4 and week 12
  Mean change in tear osmolarity from baseline as measured by Tear Lab
Change in Ocular Surface Disease Index (OSDI) score | Assessed on week 1, week 4 and week 12
  Mean change in OSDI from baseline
Change in best corrected visual acuity | Assessed on week 1, week 4 and week 12
  Mean change in Best-corrected Visual Acuity (BCVA) from baseline as measured by ETDRS chart
Physician Ease of Insertion of Dextenza | Assessed on day 1
  Physician ease of insertion as measured by a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Warrenville EyeCare & LASIK, Warrenville, Illinois, United States

IPD SHARING:
Plan to Share IPD: No